CLINICAL TRIAL: NCT04359602
Title: COVID-19 Recovered Volunteer Research Participant Pool Registry
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 20-000625
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Recovered From COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational registry of COVID-19 recovered patients who are no longer symptomatic. This Registry is intended to serve as a pool of individuals that can participate in studies associated with serological testing, characterization of immunity and immune response, vaccine development, and convalescent plasma donors.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen the in emergency room, admitted patients, or seen in outpatient clinics that are:

  * Tested Positive for COVID-19 and recovered
  * Suspected to have COVID 19 and validated with serological testing
  * Suspected to have COVID 19 by symptoms, clinical course, and laboratory testing ruling out other respiratory viral disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People volunteering to share their information to become part of this research pool of COVID-19 recovered individuals will complete an online survey.
Sampling Method: Non-Probability Sample
Enrollment: 5090 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2042-04-20 (Estimated)

PRIMARY OUTCOMES:
Serological testing of COVID patients | Up to 20 years
  Testing may be done on registry participants who agree to participate future studies
Immune response | Up to 20 years
  Testing may be done on registry participants who agree to participate future studies

CONTACTS AND LOCATIONS:
Overall Officials: Arash Naeim, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes